CLINICAL TRIAL: NCT04135950
Title: Prospective Registry of Predictors and Comorbid Injuries Associated With Anterior Cruciate Ligament Reconstructions
Brief Title: Prospective Registry of Anterior Cruciate Ligament Reconstructions
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leslie Bisson, June A. and Eugene R. Mindell, MD Professor and Chair, State University of New York at Buffalo
Other Study IDs: 441874-2
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Tear; Meniscal Tear; Cartilage Injury; Bone Bruising
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate factors that are associated with outcomes of injury to the anterior cruciate ligament (ACL) in the knee among patients who are undergoing surgical reconstruction. This study is a registry of all patients having knee surgery at our institution performed by 4 fellowship-trained orthopaedic surgeons. The surgeon documents patient information on standard data forms including risk factors and surgical findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACL surgery

Exclusion Criteria:

* Previous surgery on the affected knee
* Posterior cruciate ligament injuries
* Grade 2 lateral collateral ligament or medial collateral ligament injuries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients at our institution who are having ACL surgery by one of 4 fellowship-trained surgeons will be included in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 1646 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
additional injury | intraoperatively
  At the time of ACL surgery, it is determined if the patient has any other injuries to the meniscus or cartilage.

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Orthopaedics and Sports Medicine, Buffalo, New York, United States